CLINICAL TRIAL: NCT03183778
Title: Use of Patiromer to Transition Chronic Kidney Disease Patients With Hyperkalemia to a Plant-rich Diet.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-00051
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Results first posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Chronic Kidney Diseases; Hyperkalemia
Keywords: Chronic kidney disease, stages 3B-4
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperkalemia | interventions — patiromer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patiromer + Research Diet (Experimental): During the first phase (week 2), participants will be transitioned to a plant-rich renal diet, which contains moderate protein (10-15% of kcal), restricts dairy products (less than or equal to 1 serving/day), and eliminates high-potassium fruits and vegetables.
  During the second phase (weeks 3 and 4), the diet will be altered to provide at-least half of fruits and vegetables from high-potassium sources.
  Interventions: Drug: Patiromer; Dietary Supplement: Research Diet Menu

INTERVENTIONS:
Drug: Patiromer — Patiromer dosing will be determined based on fasting potassium concentrations measured at the end of each week, factoring in both the absolute concentration, as well as the rate of change. The baseline dose of patiromer will correspond to the study by Weir et al. (2015); 8.4-g once per day for participants with a baseline serum potassium of greater than or equal to 5.1 mEq/L.
  Other Names: Veltassa
Dietary Supplement: Research Diet Menu — During the study, participants will be asked to consume only the foods provided in the research diet

SUMMARY:
The purpose of this proof-of-concept controlled-feeding study is to determine whether patiromer (Veltassa®, Relypsa, Inc., Redwood City, CA) can be used to maintain normal serum potassium concentrations in chronic kidney disease (CKD) patients who are transitioned to a plant-rich diet.

ELIGIBILITY:
Inclusion Criteria:

* Stages 3B-4 CKD (estimated glomerular filtration rate (eGFR) of 15-44 mL/min/1.73m2, not treated with dialysis)
* No prior treatment with patiromer
* Mild hyperkalemia (potassium 5.1 to <6.5 mEq/L) on one of the last two blood tests
* No prior episodes of moderate-severe hyperkalemia (potassium ≥6.5 mEq/L) in the past 6 months
* Deemed appropriate for the intervention by the patient's nephrologist, considering the patient's prognosis, cognition and pending treatments (e.g., dialysis)

Exclusion Criteria:

* Change in medications that alter potassium homeostasis (e.g., RAAS inhibitors, diuretics, β-blockers) in the last month
* Diagnosed with bowel diseases or syndromes (e.g., bowel obstruction, major GI surgery, short-bowel syndrome, irritable bowel syndrome, inflammatory bowel disease, chronic diarrhea)
* Dietary restrictions (e.g., allergies) or otherwise unable/unwilling to adhere to study diets (excludes dietary restrictions on high-potassium foods)
* Pregnant (females) or planning to become pregnant (males and females) during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Goldfarb, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patiromer + Research Diet: During the first phase (week 2), participants will be transitioned to a plant-rich renal diet, which contains moderate protein (10-15% of kcal), restricts dairy products (less than or equal to 1 serving/day), and eliminates high-potassium fruits and vegetables.
  During the second phase (weeks 3 and 4), the diet will be altered to provide at-least half of fruits and vegetables from high-potassium sources.
  Patiromer: Patiromer dosing will be determined based on fasting potassium concentrations measured at the end of each week, factoring in both the absolute concentration, as well as the rate of change. The baseline dose of patiromer will correspond to the study by Weir et al. (2015); 8.4-g once per day for participants with a baseline serum potassium of greater than or equal to 5.1 mEq/L.
  Research Diet Menu: During the study, participants will be asked to consume only the foods provided in the research diet
Period: Overall Study
Arm/Group | Patiromer + Research Diet
Started | 3
Completed | 2
Not Completed | 1
Not completed — Withdrawn by Investigator (potassium in normal range) | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patiromer + Research Diet
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Fasting Serum Potassium Concentrations
Time Frame: Baseline, Week 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Patiromer + Research Diet
Number analyzed (Participants) | 2
mg/dL | -0.2 (0.14)

2. Primary Outcome: Change in Fasting Serum Potassium Concentrations
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Patiromer + Research Diet
Number analyzed (Participants) | 2
mg/dL | 0.7 (0.57)

3. Primary Outcome: Change in Systolic Blood Pressure (SBP)
Time Frame: Baseline, Week 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Patiromer + Research Diet
Number analyzed (Participants) | 2
mmHg | -13 (2.8)

4. Primary Outcome: Change in Systolic Blood Pressure (SBP)
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Patiromer + Research Diet
Number analyzed (Participants) | 2
mmHg | -14.9 (11.9)

5. Primary Outcome: Change in Diastolic Blood Pressure (DBP)
Time Frame: Baseline, Week 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Patiromer + Research Diet
Number analyzed (Participants) | 2
mmHg | -5.5 (2.1)

6. Primary Outcome: Change in Diastolic Blood Pressure (DBP)
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Patiromer + Research Diet
Number analyzed (Participants) | 2
mmHg | -4.3 (4)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Patiromer + Research Diet
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT03183778/Prot_SAP_000.pdf